CLINICAL TRIAL: NCT03442894
Title: Dry Needling in Addition to Standard Physical Therapy Treatment for Sub-Acromial Pain Syndrome: A Randomized Controlled Trial
Brief Title: Dry Needling for Sub Acromial Pain Syndrome
Acronym: DITTO SAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Benjamin Hando, Orthopedic and Rehabilitation Flight Commander, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20170083H
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Shoulder pain; Subacromial; bursitis; rotator cuff; tendinopathy; dry needling; myofascial trigger point
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Bursitis; Tendinopathy | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: 3 groups: Standard physical therapy treatment (SPT), SPT plus dry needling and SPT plus sham dry needling
Who Masked: Participant
Masking Description: Subjects in the dry needling and sham dry needling groups will be masked (blinded) to whether or not they are receiving the sham or actual dry needling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard PT Treatment (Active Comparator): This group will receive manual therapy and exercise interventions provided by their physical therapist. The treatment will occur for 10 sessions over 6 weeks.
  Interventions: Manual therapy interventions including mobilization and manipulation of the shoulder girdle spine and ribcage. Exercise interventions will include strengthening and flexibility exercises for rotator cuff and shoulder girdle musculature.
  Interventions: Procedure: Standard Physical Therapy Treatment
- Standard PT Treatment plus DN (Experimental): In addition to the standard PT interventions, the Dry Needling (DN) group will receive 6 DN sessions as part of their rehabilitation visits.
  Interventions: Procedure: Standard Physical Therapy Treatment; Procedure: Dry Needling
- Standard PT Treatment plus Sham DN (Sham Comparator): In addition to the standard PT treatment, patients in the sham DN group will receive 6 sessions of sham DN intervention.
  Interventions: Procedure: Standard Physical Therapy Treatment; Procedure: Sham Dry Needling

INTERVENTIONS:
Procedure: Standard Physical Therapy Treatment — All three groups will receive manual therapy and exercise interventions provided by their physical therapist. The exact dosage and choice of exercise and manual therapy techniques will not controlled in the study. Documentation of dosage and utilization rates of each will be captured for each patient session in order to determine if these variables influence outcomes. A full shoulder exam will be conducted per standard of care at this time as well. Manual therapy and exercise interventions will be selected to address impairments uncovered in the shoulder exam.
Procedure: Dry Needling — In addition to the standard PT interventions, the Dry Needling (DN) group will receive 6 DN sessions as part of their rehabilitation visits (they will occur at the same time). In 6 of the scheduled 10 visits, dry-needling intervention will be performed. They will have one DN session per week, which is consistent with typical clinical practice. After they complete their standard PT treatment, and while still in the clinic, the rotator cuff and periscapular muscles will be evaluated for the presence of MTrPs. Once located, the MTrPs will be treated with DN technique, as this is consistent with routine clinical practice. Potential muscles to receive TPDN treatment include the following: suprapsinatus, teres minor, infraspinatus, deltoid, upper trapezius, middle trapezius, levator scapula, pec major and pec minor.
  Arms: Standard PT Treatment plus DN
Procedure: Sham Dry Needling — In addition to the standard PT treatment, patients in the sham DN group will receive what appears to be a DN treatment, but it will not be done with the acupuncture needles and the skin will not be punctured. The Sham DN procedure will be performed over the site of identified MTrPs using a guide tube and a toothpick. A guide tube is positioned firmly over the area to be treated and a toothpick is inserted in the guide tube. The clinician taps the toothpick to mimic the skin prick from a needle and the guide tube is removed. The clinician maintains pressure on the end of the toothpick and moves the end furthest from the skin in different directions to mimic the pistoning and changes in needle angle that occur in actual dry needling. Care will be taken to treat from 1-3 muscle groups for 5-10 seconds per MrTP identified.
  Arms: Standard PT Treatment plus Sham DN

SUMMARY:
This trial will investigate the benefit of trigger point dry needling (DN) for individuals with a common cause of shoulder pain - sub-acromial pain syndrome. Sub-acromial pain syndrome, also knowns as SAPS, is one of the most common causes of shoulder pain. Physical therapy treatments are routinely used for treating SAPS. One treatment approach that has been shown to be beneficial is a combination of exercises and manual or manipulative therapy. This approach has been shown to reduce pain and improve overall shoulder function in individuals with SAPS.

Recently, a novel treatment approach for SAPS has emerged that involves trigger point DN to muscles of the shoulder and ribcage. Some studies have shown promising results for this approach while others have not found it to be helpful. Overall there is currently little research available on the benefit of trigger point DN for individuals with SAPS.

This study will investigate whether adding trigger point DN to a treatment program of exercise and manual therapy provides any benefit to individuals with SAPS. To answer this question, this study will divide subjects into three groups. One group will receive just exercise and manual therapy; one group will receive manual therapy and exercise plus trigger point DN and one group will receive manual therapy and exercise plus a sham trigger point DN treatment.

All patients receiving treatment in the study will attend 10 visits to a physical therapy clinic over a 6-week period. Subjects in the dry needling and sham dry needling groups will receive 6 sessions of this treatment in addition to their 10 sessions of exercise and manual therapy.

The investigators will assess the effectiveness of the three treatment protocols by measuring patients pain, shoulder function and disability levels. These outcomes will be assessed at baseline, six weeks, 6 months and one year from enrolling in the study.

In addition to assessing clinical outcomes following treatment, the investigators will assess the amount of health care utilized by each participant in the year following enrollment in the study. The 3 groups will be analyzed to determine if there is a difference in the amount or type of additional healthcare utilized in the year following study enrollment. Examples of healthcare utilization include x-rays, medication and/or surgical procedures.

The investigators hypothesis is that individuals that receive actual trigger point DN in addition to manual therapy and exercise interventions will demonstrate greater improvements in pain, shoulder function and disability when compared to individuals receiving exercise and manual therapy alone or exercise and manual therapy with sham needling. The investigators think these differences in clinical outcomes will be present at each of the follow-up points. Additionally, the investigators hypothesize that individuals receiving actual DN will use less healthcare than those in the other two groups.

DETAILED DESCRIPTION:
STUDY PURPOSE:

The purpose of this study is to assess the long-term additive effectiveness of dry needling (DN) therapy to a standard physical therapy (PT) approach of manual therapy and exercise for patients with subacromial pain syndrome.

HYPOTHESIS AND PRIMARY AIM:

Primary Aim: Compare 1-year outcomes in patients that receive standard PT treatment versus standard PT and DN versus standard PT and sham DN, in patients with SAPS (self-reported outcomes and shoulder-related healthcare utilization). Standard PT will consist of therapeutic exercise and manual therapy, which is considered standard of care PT treatment for individuals with SAPS.

The hypothesis for the primary aim: DN in addition to standard PT treatment will be more effective than standard PT alone. There will be no difference between the Sham DN + standard PT and the standard PT only groups.

BACKGROUND AND SIGNIFICANCE:

Subacromial pain syndrome (SAPS) is among the most common and self-limiting disorders of the musculoskeletal system. The point prevalence of shoulder symptoms has been reported to range from 20-33% and the incidence of shoulder complaints in the general population is increasing. Furthermore, several authors have reported low rates of perceived recovery (patient reports of "being cured") for patients with a new episode of shoulder or neck pain. According to Bot et al, less than 25% of patients with a first episode of shoulder pain reported recovery after 3 months, and only 32% stated they had recovered (no longer had symptoms) after 1 year. Other studies have investigated the prognosis of shoulder pain in general practice. Pope et al reported recovery rates of only 21% after 6 months and 49% after 18 months. Van der Windt et al and Winters et al reported recovery rates of 51% and 59% after 12 to 18 months, respectively. Finally, Rekola et al reported that 25% of patients with shoulder or neck pain experienced at least one episode of recurrence within 12 months. These findings suggest that shoulder pain can be recurrent and frequently progresses to the chronic stage. This is clearly a musculoskeletal condition requiring further research to identify effective management strategies.

RESEARCH DESIGN AND METHODS:

This will be a randomized clinical trial with 3 arms. This is a pragmatic comparative effectiveness trial utilizing interventions that are all standard of care and already utilized in clinical care. The experimental nature of the study is the comparative effectiveness using sham needling, and the assessment of whether an additive combination of treatments is better than the standard treatment alone.

Self-reported outcome measures will be captured at baseline, 6 weeks, 6 months, and 1 year. The investigators will observe healthcare-related expenditures and utilization for all groups for one year following enrollment in order to uncover differences in health-seeking behaviors and health care cost following the intervention between the treatment groups.

INTERVENTIONS:

Randomization: Subjects will then be randomized into one of three arms (Group I = Standard PT Treatment PLUS TPDN, Group II = Standard PT Treatment PLUS Sham TPDN, Group III = Standard PT Treatment only). The method of group assignment will be sequentially numbered opaque sealed envelopes (SNOSE). To minimize the risk of predicting the treatment assignment of the next eligible patient, randomization will be performed in permuted blocks of 2 or 4 with random variation of the blocking number. All self-report measures will be filled out prior to randomization.

Blinding: Due to the nature of this study, it is not possible to fully blind the patient or the clinician providing the intervention to the treatment received, although the patient will not know the details of the other study groups in which they are not a part of. The patient will be blinded to whether they receive real or sham TPDN, but they will know if they are in the group does not receive either. The evaluator and physical therapist providing the intervention will be different individuals. The assessor performing the baseline measurements and outcome assessments will be blinded to the patient's group assignment. Patients will be instructed not to discuss the intervention received with the assessor unless medically necessary. Incidence of unmasking will be recorded.

Treatment Groups Description:

This will be a pragmatic study, where patients will be required to try and attend at least 10 sessions over a 6-week period, but can attend more if the therapist believes there is still progress to be made. This mimics actual clinical practice. The number of actual sessions will be recorded.

Standard PT Treatment: All three groups will receive manual therapy and exercise interventions provided by their physical therapist. The exact dosage and choice of exercise and manual therapy techniques will not controlled in the study. Documentation of dosage and utilization rates of each will be captured for each patient session in order to determine if these variables influence outcomes. A full shoulder exam will be conducted per standard of care at this time as well. All treating clinicians will receive a basic training session to review the exercise and manual therapy techniques that will be used.

Dry Needling:

In addition to the standard PT interventions, the Dry Needling (DN) group will receive 6 DN sessions as part of their rehabilitation visits (they will occur at the same time). In 6 of the scheduled 10 visits, dry-needling intervention will be performed. They will have one DN session per week, which is consistent with typical clinical practice. After they complete their standard PT treatment, and while still in the clinic, the rotator cuff and periscapular muscles will be evaluated for the presence of MTrPs. Once located, the MTrPs will be treated with DN technique, as this is consistent with routine clinical practice. Potential muscles to receive TPDN treatment include the following: suprapsinatus, teres minor, infraspinatus, deltoid, upper trapezius, middle trapezius, levator scapula, pec major and pec minor.

SEIRIN Acupuncture needles (50mm length; 0.30mm diameter) will be used to perform the dry needling procedure. The skin will be prepped with an alcohol swab, gloves will be worn and clean needle technique will be used at all times. The needle will be inserted over the MTrP with a goal of inserting to the depth of the MTrP in an attempt to elicit a local twitch response (LTR). After needle insertion the treating clinician will "piston" the needle (in and out motion). Pistoning will be performed for approximately 5-10 seconds. Each MTrP will be treated in this fashion with up to 3 muscle groups treated within a single session. Clinicians will document the location of MTrP's and at which visit they were identified and treated.

Sham DN: In addition to the standard PT treatment, patients in the sham DN group will receive what appears to be a DN treatment, but it will not be done with the acupuncture needles and the skin will not be punctured. The Sham DN procedure will be performed over the site of identified MTrPs using a guide tube and a toothpick. The clinician preps the skin with an alcohol wipe and holds the skin taut around the area in contact with the needle, just as is done in actual dry-needling technique. A guide tube is positioned firmly over the area to be treated and a toothpick is inserted in the guide tube. The clinician taps the toothpick to mimic the skin prick from a needle and the guide tube is removed. The clinician maintains pressure on the end of the toothpick and moves the end furthest from the skin in different directions to mimic the pistoning and changes in needle angle that occur in actual dry needling. Care will be taken to treat from 1-3 muscle groups for 5-10 seconds per MrTP identified. Following completion of the 6-week treatment period, subjects will be asked to identify which treatment group they were it in order to assess if the sham procedure was successful in mimicking the DN procedure.

SETTING:

This study will take place in the physical therapy clinics at Wilford Hall Ambulatory Surgical Center (WHASC), on Lackland Air Force Base in San Antonio, TX and the CPT Jennifer Moreno PT clinic at Fort Sam Houston, San Antonio TX.

RISK:

As with all clinical research, there is a small risk of inadvertent breach of confidentiality of PHI/PII. The likelihood of this breach is low given the efforts the research team will take to protect this information.

Potential risks to subjects in this study are minimal. The procedures used in this study are standard procedures that are used in everyday clinical practice in the PT clinics that are participating. The use of manual therapy and exercise treatments for patients with subacromial pain syndrome is supported by clinical practice guidelines in the United States and elsewhere. There are no associated study-related risks with the treatment, as it is all standard of care. Although there are no research-related risks associated with this study, there are some minor risks from the procedures used in this study, which would be present regardless of whether the patient decides to participate in the study or not. If they participate in physical therapy, there is a risk for increased pain or muscle soreness as a result from exercise and manual therapy procedures used in physical therapy. The majority of these instances are transient, lasting less than 24 hours.

The risks from the DN needling intervention are also minor and transient. Specifically, there is a small risk of pain, bruising and bleeding. The likelihood of these occurrences is approximately 20%. They are characterized as minor because they resolve within 24 hours and do not require additional medical attention. There is a small risk of more serious medical events with dry needling. These include haematoma, pneumothorax, and nerve lesion. These occurrences are very rare, occurring at a rate of < 0.04%.50

Although the risks to patients related directly to the study are extremely low, the investigators will implement monitoring procedures to ensure the safety and protection of subjects. Members of the research team are credentialed providers, and familiar with managing patients with shoulder pain. The research team will always monitor the safety and appropriateness of each patient in the study. All personnel involved with the research who will be responsible for collecting and handling the data will have completed the CITI training and will be trained by one of the investigators. Protection of patient confidentiality and procedures for reporting adverse events will be included in these training sessions. Any adverse events occurring as a result of participation in this study will be reported immediately to the principal investigator and the Institutional Review Board involved with the study. The Principal Investigator will meet on a weekly basis with the study staff to review study progress, including any adverse events or breaches of patient confidentiality.

DATA ANALYSIS All data will be analysed in IBM SPSS 24 (Chicago, IL). Descriptive statistics will be performed to describe the sociodemographic (age, sex, race, etc.) and health characteristics (disability, pain intensity, psychosocial factors, etc.) of the entire sample, and comparisons made between groups. Means and standard deviations will be computed for continuous data and frequency distributions will be analyzed for categorical data. For differences in shoulder-related healthcare utilization, RRs (risk ratio) for a healthcare utilization event between patients in each group will be derived and compared. Point estimates with 95% Confidence Intervals will be reported.

Comparison of self-report outcomes between groups at baseline, 6 weeks, 6 months and 1 year will be performed using a linear mixed-effects model, which is flexible in accommodating data assumed to be missing at random. Significance is set at 0.05 and 95% confidence intervals will be reported for all relevant data. Sensitivity analysis will be run adjusting for other demographic and/or prognostic variables (OSPRO-YF, pain intensity, PROMIS-29 sleep or mental health domains, etc) that may affect the outcome.

Sample Size: In order to generate 80% power for this study, with 3 potential treatment arms, based an effect size difference in SPADI scores of 12%, the investigaros need a total sample size of 108 subjects (36 per group). With an estimated 20% loss to follow-up or drop outs at 1 year, the investigators will plan on enrolling 130 subjects into the study in order to have 108 complete their 1-year follow-ups. Calculations derived with G*Power.

FUNDING SUPPORT: None

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Read and speak English well enough to provide informed consent, follow study instructions, and independently answer the questionnaires/surveys
* Tricare beneficiary
* Primary complaint of new episode of shoulder pain; defined as not having sought care for shoulder condition in 6 months prior
* Available and willing to come in for treatment (~10 sessions over 6 week period)
* Meets criteria for SAPS from description below, by having 2 of the 4 following physical exam findings:
* Impingement signs (Neer, Hawkins, or Jobe tests)
* Painful arc
* Pain with isometric resistance (ER/IR/ABD)
* Rotator cuff weakness on the injured side in comparison to the opposite side

Exclusion Criteria:

* History of shoulder dislocation, subluxation, fracture, adhesive capsulitis of the glenohumeral joint, or cervical/shoulder/upper back surgery
* Presence of cervical radiculopathy, radiculitis, or referral from cervical spine
* Total baseline SPADI score less than 20% (to prevent a ceiling effect with treatment)
* Anyone pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury
* Unable to give informed consent to participate in the study.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) scores | Baseline, 6-weeks, 6 months, 12 months
  The SPADI is a 100-point, 13 item self-administered questionnaire. It is divided into two subscales: a five item pain subscale and an eight-item disability subscale. Williams et al have shown that the SPADI is responsive to change and accurately discriminates between patients who are improving or worsening. Michener and Leggin also reported a high test-retest reliability and internal consistency for this instrument. When compared to the Sickness Impact Profile (SIP), Heald et al found that the construct validity of the SPADI is moderately strong and it is more responsive to change than the SIP. A recent systematic review identified a minimal detectable change (MDC) of 18 and a minimally clinically important difference (MCID) of between 8-13 points. The validity and responsiveness to change of SPADI have been described in physical therapy, as well as primary and secondary care settings.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information Systems (Promis-29) | Baseline, 6 weeks, 6 months, 12 months
  The Patient-Reported Outcomes Measurement Information Systems (PROMIS) 29-item short form (version 2). The PROMIS 29-item short form efficiently assesses several outcomes important to patients; including, pain intensity and interference, sleep disturbance, anxiety, depression, fatigue, and social role participation using items developed with rigorous methodology and patient input.
Patient Acceptable Symptom Scale (PASS) | Baseline, 6 weeks, 6 months, 12 months
  Often defined as "the highest level of symptoms beyond which patients consider themselves well." This outcome measure has been used in previous studies looking at the effects of cervico-thoracic thrust manipulation on shoulder pain. The question that will be asked to assess this level is, "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" Individuals who responded "yes" were categorized as a success." Between group differences at four time points will be assessed as percentage of subjects who find their current state acceptable, or answering "yes."
Optimal Screening for Prediction of Referral and Outcome Yellow Flags assessment tool (OSPRO-YF) | Baseline, 6 weeks, 6 months, 12 months
  The OSPRO-YF measures psychosocial risk factors. It may be administered early after injury and sequentially over time.
Healthcare Utilization | 12 months following enrollment
  Healthcare utilization data will be collected from the Military Health System (MHS) Data Repository (MDR) database. Healthcare utilization data will be used to determine any subsequent medical utilization related to shoulder pain. The goal of the MDR database will be to determine which of these subjects sought health care related to shoulder pain in the 12-month period after treatment in this study. This data (type, location, number of clinic visits, types of specialty clinic visits, imaging, and associated medication) will allow us to determine the extent of healthcare utilizations incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Hando, DScPT, Principal Investigator — US Air Force
Locations (1):
- Wilford Hall Ambulatory Surgical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share the data with other researchers. Our team has not coordinated with other researchers to share our data.

REFERENCES:
- [Background] Rhon DI, Boyles RB, Cleland JA. One-year outcome of subacromial corticosteroid injection compared with manual physical therapy for the management of the unilateral shoulder impingement syndrome: a pragmatic randomized trial. Ann Intern Med. 2014 Aug 5;161(3):161-9. doi: 10.7326/M13-2199. PMID 25089860
- [Background] Pope DP, Croft PR, Pritchard CM, Silman AJ. Prevalence of shoulder pain in the community: the influence of case definition. Ann Rheum Dis. 1997 May;56(5):308-12. doi: 10.1136/ard.56.5.308. PMID 9175931
- [Background] Perez-Palomares S, Olivan-Blazquez B, Perez-Palomares A, Gaspar-Calvo E, Perez-Benito M, Lopez-Lapena E, de la Torre-Beldarrain ML, Magallon-Botaya R. Contribution of Dry Needling to Individualized Physical Therapy Treatment of Shoulder Pain: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2017 Jan;47(1):11-20. doi: 10.2519/jospt.2017.6698. Epub 2016 Dec 10. PMID 27937046
- [Background] Koppenhaver S, Embry R, Ciccarello J, Waltrip J, Pike R, Walker M, Fernandez-de-Las-Penas C, Croy T, Flynn T. Effects of dry needling to the symptomatic versus control shoulder in patients with unilateral subacromial pain syndrome. Man Ther. 2016 Dec;26:62-69. doi: 10.1016/j.math.2016.07.009. Epub 2016 Jul 21. PMID 27497188
- [Derived] Hando BR, Rhon DI, Cleland JA, Snodgrass SJ. Dry needling in addition to standard physical therapy treatment for sub-acromial pain syndrome: a randomized controlled trial protocol. Braz J Phys Ther. 2019 Jul-Aug;23(4):355-363. doi: 10.1016/j.bjpt.2018.10.010. Epub 2018 Nov 6. PMID 30455091